CLINICAL TRIAL: NCT01822717
Title: Nonvisual Foot Inspection for People With Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Kent State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BRIDGES- ST09 49
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes; Visual Impairment
Keywords: Diabetes; Visual Impairment; Blindness; Foot Care; Self-Management
MeSH Terms: conditions — Diabetes Mellitus; Vision Disorders; Blindness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nonvisual foot inspection (Experimental): Instruction for nonvisual foot inspection included in comprehensive diabetes self-management education
  Interventions: Behavioral: Nonvisual foot inspection
- Usual Care for foot inspection (Active Comparator): Usual instruction for foot care included in comprehensive diabetes self-management education
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Nonvisual foot inspection — Teaching use of nonvisual senses (tactile and olfactory) to empower people with diabetes and visual impairment to perform a systematic self-examination of their own feet
  Other Names: Multi-SAFE (Multiple Senses And Foot Examination)
  Arms: Nonvisual foot inspection
Behavioral: Usual Care — Standard instructions for foot care for people with visual impairment include advice to have a sighted family member or friend check the person's feet regularly
  Other Names: Standard foot care instructions
  Arms: Usual Care for foot inspection

SUMMARY:
The purpose of this study was to find out whether a method of nonvisual foot inspection, using the senses of touch and smell, helps people with diabetes and visual impairment to find new foot problems when they are in early, easily-treated stages. All people in the study had regular foot inspections by podiatrists. The results include how people feel about the method, whether they actually did check their feet it, and whether the method helped them to discover foot problems themselves.

DETAILED DESCRIPTION:
Data gathered over the course of 1 year:

* bimonthly phone calls to ask about foot care practices at home over the last week
* a baseline comprehensive foot evaluation and 4 additional comprehensive evaluations every 3 months

Qualitative data:

- Focus groups immediately after comprehensive diabetes self-management education, and 1 year later, to determine acceptability of foot care procedures and patient perceptions about effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Diagnosed with diabetes (either type 1 or type 2)
* Having visual impairment

Exclusion Criteria:

* Self-reported numbness in hands
* Inability to pass a brief screening for decisional capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Days per week participants performed foot inspection | every 2 months for 1 year
  Number of days in the last week each participants reported checking their feet for problems, using nonvisual methods (experimental group) or with assistance form someone else (comparison group)

SECONDARY OUTCOMES:
Number of foot problems discovered | every 3 months for 1 year
  Number of foot problems discovered by podiatrists or at home by participants

OTHER OUTCOMES:
Acceptability | 1 year
  Qualitative information from focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Ann S Williams, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Cleveland Foot and Ankle Institute, Cleveland, Ohio, United States

REFERENCES:
- [Background] Williams A. Appraising the Multi-SAFE approach to low vision and diabetes: a simple technique for saving feet. Diabetes Voice 56(Special Issue 1):14-17, 2011